CLINICAL TRIAL: NCT06368011
Title: The Effect of Acceptance and Commitment Therapy-Based Psychoeducation on Stigmatization Levels of Schizophrenia Patient Relatives
Brief Title: The Impact of Acceptance and Commitment Therapy on Stigmatization
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mustafa Kemal University (Other)
Responsible Party: Principal Investigator, Gamze Cincinoglu, teaching assistant, Mustafa Kemal University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: MustafaKU-CINCINOGLU-001
Record Dates: First submitted 2024-03-18; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Stigmatization
Keywords: acceptance and commitment therapy; schizophrenia; family; stigma
MeSH Terms: conditions — Stereotyping; Schizophrenia; Social Stigma | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group:relatives of schizophrenia patients (Experimental): The population of the study consisted of the relatives of schizophrenia patients who were registered and actively attending the Ministry of Health Dr. Nafiz Körez Sincan State Hospital Community Mental Health Center.The sample size of the study was calculated at 95% confidence level according to the independent t test using 'G. Power-3.1.9.7' before the study was started.As a result of the analysis, the minimum sample size was calculated as 32, with 16 in the experimental group and 16 in the control group.
  Interventions: Behavioral: acceptance and commitment therapy
- control group:relatives of schizophrenia patients (No Intervention)

INTERVENTIONS:
Behavioral: acceptance and commitment therapy — Psychoeducation was delivered in 8 sessions lasting 90 minutes to two separate groups of 8-10 individuals in the experimental group.Group sessions were conducted once a week at the community mental health center under the leadership of the researcher.In total, the psychoeducation lasted 10 weeks, including make-up sessions.
  Arms: experimental group:relatives of schizophrenia patients

SUMMARY:
The goal of study is to determine the effect of acceptance and commitment therapy-based psychoeducation on the level of stigmatization applied to relatives of schizophrenia patients.

Type of study: This study was planned as a pretest-posttest quasi-experimental design with an observation and control group.

Participants: The population of the study consisted of the relatives of schizophrenia patients who were registered and actively attending the Community Mental Health Center in a state hospital in Ankara.

Intervention: Before the psychoeducation process started, personal information form and scales were applied to the relatives of the patients in the experimental and control groups. An ACT-based psychoeducation program consisting of 8 sessions was applied to the experimental group. each session lasted approximately 90 minutes. The control group did not receive any intervention. After the psychoeducation, the scales were reapplied to the experimental and control groups. In addition, the experimental group was asked to fill out the psychoeducation evaluation form. The scales were reapplied to the experimental group after the 1-month follow-up study and evaluated.

DETAILED DESCRIPTION:
Aim The aim of this study is to determine the effect of Acceptance and Commitment Therapy (ACT)-based psychoeducation on the level of stigmatization of mental illness in the relatives of individuals diagnosed with schizophrenia.

Study Desing The design of the study is an experimental research with pretest-posttest, follow-up measurement experiment and control group.

Hypotheses The reserach hypotheses are as follows; H0: acceptance and commitment therapy has no effect on the level of stigmatization.

H1: Psychoeducation based on acceptance and commitment therapy is effective in reducing the stigmatization levels of relatives of schizophrenia patients.

Variables of the study The study's dependent variable is stigma , and the independent variable is ACT based psychoeducation.

Settings The research was conducted between April 2023 and July 2023 with the relatives of patients diagnosed with schizophrenia who were followed up at the Ministry of Health Dr. Nafiz Körez Sincan State Hospital Community Mental Health Center.

Participants The sample of this study consisted of relatives of patients diagnosed with schizophrenia who were followed up in Dr. Nafiz Körez Sincan State Hospital Community Mental Health Center. After determining the sufficient number of relatives for the sample, randomization was performed. The relatives of the patients included in the study were randomly assigned to the experimental and control groups. There was no loss of sample in both groups during the psychoeducation period and the study was completed with 36 relatives of the patients.

Information Form: the researcher prepared this form, consisting of questions about the sociodemographic characteristics of relatives of schizophrenia patients, stigmatization scale and stigma scale for relatives of schizophrenia patients.

Stigma Scale For Relatives of Schizophrenia Patients.The scale developed by Yıldırım et al. was prepared as a 3-point Likert-type scale. Yes: 3, Sometimes: 2, No: 1 and scored as Yes: 3, Sometimes: 2, No: 1. The minimum score that can be obtained from the scale is 17 and the maximum score is 51. There are no reverse scored items. The scale is interpreted on both the total score and the subscale scores, and the higher the score obtained from the scale and subscales, the more stigmatization is expressed. The stigmatization scale for relatives of schizophrenia patients consists of 17 questions and 5 subscales. Social isolation and inadequacy sub-dimension 1, 2, 3, 4, 9, 15 avoidance and deterioration in interpersonal relationships sub-dimension: 5, 6, 7 social negative discrimination sub-dimension: 8, 10, 11 concealment and shame subscale: 12, 13, 14 negative internalization subscale: 16, 17 items. In the reliability study, the Cronbach's Alpha coefficient of the scale was found to be 0.90. The Cronbach's Alpha internal consistency coefficients of the Stigma Scale for Relatives of Schizophrenia Patients were calculated as 0.87; 0.80; 0.76; 0.71; 0.69 for the sub-dimensions of social isolation and inadequacy, avoidance and deterioration in interpersonal relationships, social negative discrimination, concealment and shame, and negative internalization, respectively. In the present study, the reliability of the CCPBS scale was found to be high as Cronbach's Alpha=0.839.

Stigmatization Scale: The scale is a 5-point Likert-type. It is answered and scored as Strongly Disagree: 1, Disagree: 2, Partially Agree: 3, Agree: 4, Strongly Agree: 5. The score that can be obtained from the scale is between 22-110, and it can be said that individuals who score below 55 points have a low stigmatization tendency, while individuals who score above 55 points have a high stigmatization tendency. The Stigmatization Scale consists of 22 items and 4 dimensions and there are no reverse scored items. Discrimination and exclusion sub-dimension 10,17,18,19,20,21 labeling sub-dimension 3,4,5,7,8,9 psychological health sub-dimension 11,12,13,15,16, prejudice sub-dimension 1,2,6,14,22. In the reliability study, Cronbach's Alpha coefficient of the scale was found to be 0.84. Cronbach's Alpha internal consistency coefficients of the Stigma Scale were found to be 0.77, 0.68, 0.66, 0.54 for discrimination and exclusion, labeling, psychological health, and prejudice sub-dimensions, respectively. In this study, the reliability of the Stigmatization scale was found to be high as Cronbach's Alpha=0.827.

Data Collection: Before the psychoeducation process started, personal information form and scales were applied to the relatives of the patients in the experimental and control groups. ACT-based psychoeducation program was applied to the experimental group. The psychoeducation program was carried out in 8 sessions, each session lasting approximately 90 minutes. The control group did not receive any intervention. After the psychoeducation program given to the experimental group, the scales were reapplied to the experimental and control groups. In addition, the experimental group was asked to fill out the psychoeducation evaluation form. After 1 month of follow-up study, the scales were applied to the experimental group again and evaluated.

Psychoeducation was provided to two separate groups of 8-10 individuals in the experimental group in 8 sessions lasting 90 minutes. The group sessions were conducted once a week at the TRSM under the leadership of the researcher. In total, the psychoeducation lasted 10 weeks including make-up sessions. The sessions were held in the multi-purpose training hall of the TRSM, which had appropriate conditions for psychoeducation (a table and enough chairs, blackboard, computer, overhead projector).

Data Analysis The data obtained in the study were evaluated in computer environment through SPSS 22.0 statistical program. Frequency and percentage analyses were used to determine the descriptive characteristics of the employees participating in the study, and mean and standard deviation statistics were used to examine the scale. Kurtosis and Skewness values were analyzed to determine whether the research variables were normally distributed. It was determined that the variables were normally distributed. Parametric methods were used to analyze the data.Differences between the rates of categorical variables in independent groups were analyzed with Chi-Square and Fisher exact tests. Independent groups t-test was used to compare quantitative continuous data between two independent groups. Repeated measures anova test and complementary bonferroni test were used to compare within-group measurements.

Funding No expenditure will be made on any item other than the consumables of the existing forms for the research. the researcher will cover stationery and consumables.

ELIGIBILITY:
Inclusion Criteria:

* Being a relative of a patient diagnosed with schizophrenia according to DSM-V diagnostic criteria
* Living with the patient (family member living with the patient for at least 35 hours or more per week)
* Volunteering to participate in the research,
* To be able to read and write
* 18 years of age or older

Exclusion Criteria:

* Not having attended any session of the eight-session training program and not having attended the make-up session
* Not having participated in any of the pre-test, post-test and follow-up test

Min Age: 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-04-15 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Stigma Scale for Relatives of Patients with Schizophrenia | Pre-test (before the intervention), post test (ten weeks after the intervention) and one month after follow up
  It is a 3-point Likert-type scale. Yes: 3, Sometimes: 2, No: 1 and is scored as followsThe lowest score that can be obtained from the scale is 17 and the highest score is 51.
Stigma Scale for Relatives of Patients with Schizophrenia | post test (ten weeks after the intervention)
  It is a 3-point Likert-type scale. Yes: 3, Sometimes: 2, No: 1 and is scored as followsThe lowest score that can be obtained from the scale is 17 and the highest score is 51.
Stigma Scale for Relatives of Patients with Schizophrenia | one month after follow up
  It is a 3-point Likert-type scale. Yes: 3, Sometimes: 2, No: 1 and is scored as followsThe lowest score that can be obtained from the scale is 17 and the highest score is 51.

SECONDARY OUTCOMES:
Stigmatization Scale | Pre-test (before the intervention), post test (ten weeks after the intervention) and one month after follow up
  It is a 5-point Likert-type scale. It is answered and scored as Strongly Disagree: 1, Disagree: 2, Partially Agree: 3, Agree: 4, Strongly Agree: 5. The score that can be obtained from the scale is between 22-110, and it can be said that individuals who score below 55 points have a low tendency to stigmatize, while individuals who score above 55 points have a high tendency to stigmatize.
Stigmatization Scale | post test (ten weeks after the intervention)
  It is a 5-point Likert-type scale. It is answered and scored as Strongly Disagree: 1, Disagree: 2, Partially Agree: 3, Agree: 4, Strongly Agree: 5. The score that can be obtained from the scale is between 22-110, and it can be said that individuals who score below 55 points have a low tendency to stigmatize, while individuals who score above 55 points have a high tendency to stigmatize.
Stigmatization Scale | one month after follow up
  It is a 5-point Likert-type scale. It is answered and scored as Strongly Disagree: 1, Disagree: 2, Partially Agree: 3, Agree: 4, Strongly Agree: 5. The score that can be obtained from the scale is between 22-110, and it can be said that individuals who score below 55 points have a low tendency to stigmatize, while individuals who score above 55 points have a high tendency to stigmatize.

CONTACTS AND LOCATIONS:
Locations (1):
- Hatay Mustafa Kemal Üniversitesi, Hatay, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Pre-test and post-test scores of relatives of schizophrenia patients will be matched with coding. relatives of schizophrenia patients will be asked to code the codes consisting of the first letter of their surname, the last two digits of their